CLINICAL TRIAL: NCT06758661
Title: An Open-label, Single-arm, Crossover, Multiple-dose Phase 1 Study to Evaluate Drug-drug Interaction and Safety After the Co-administration of D352 and D794, in Healthy Adult Volunteers
Brief Title: Clinical Study to Evaluate Drug-drug Interaction and Safety After Co-administration of D352 and D794 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A149_01DDI2409
Record Dates: First submitted 2024-12-26; First posted 2025-01-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — 1-stearoyl-d35-2-docosahexaenoyl-sn-glycero-3-phosphocholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D352-D352+D794(Part 1) (Experimental): Period 1: D352 1 tablet for 1 week, Period 2: D352 1 tablet and D794 4 capsule for 2 weeks
  Interventions: Drug: D352; Drug: D794
- D794-D352+D794(Part 2) (Experimental): Period 1: D794 4 capsule for 2 weeks, Period 2: D352 1 tablet and D794 4 capsule for 1 week
  Interventions: Drug: D352; Drug: D794

INTERVENTIONS:
Drug: D352 — 1 tablet
Drug: D794 — 4 capsule

SUMMARY:
This study is a randomized, open-label, single arm, multi-dose, crossover study to evaluate drug-drug interaction and safety after co-administration of D352 and D794 in healthy adult volunteers.

DETAILED DESCRIPTION:
36 healthy subjects are administration of D352 and D794 following each part. Pharmacokinetic blood samples are collected 1d to 22d. The drug-drug interaction and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers between the ages of 19 years to 55 years.
2. Individuals who had 18 kg/m2 ≤ Body Mass Index(BMI) < 30 kg/m2 and total body weight ≥ 55 kg (woman total body weight ≥ 45 kg) BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination
4. Individuals who were deemed to be appropriate as study subjects following vital sign, laboratory tests (hematology, blood chemistry, serology, urology etc.) etc. performed
5. Individuals who agreed proper contraception during the study and did consent to not donation of sperm or eggs 14 days after the last dose of study drug
6. Individuals who signed an informed consent form after being fully informed of the study prior to participation, including the objective, content, adverse events etc.

Exclusion Criteria:

1. Individuals with a history of hypersensitivity to any of the major ingredients or components of the investigational product
2. Individuals who have genetic problems such as galactose intolerance, Lap lactase deficiency, or glucose-galactose malabsorption
3. Individuals who have a history of hypersensitivity or allergy to this ingredient because it contains Sunset Yellow FCF
4. Patients with the following diseases

   * Patients with active liver disease or persistently elevated aminotransferase levels of unknown cause
   * Patients with severe hepatic impairment of biliary obstruction and patients with cholestasis
   * Patients receiving cyclosporine
   * Myopathic patients
5. Individuals with a history of gastrointestinal surgery or gastrointestinal disease that may affect drug absorption
6. Individuals who exceed the following condition with 1 month of the first administration of investigational product

   * Alcohol: Man-21 glasses/week, Woman-14 glasses/week (1 glass = soju 50mL or liquor 30mL or beer 250mL)
   * Smoking: 20 cigarettes/day
7. Individuals who cannot restrict the intake of grapefruit or food containing grapefruit from three days before the first administration of investigational product until the final pharmacokinetic blood sample is collected
8. Individuals who have used drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the first dosing administration
9. Individuals who have taken any specialty or herbal medicine within 2 weeks prior to the first administration, or any over-the-counter(OTC) or dietary supplement or vitamin preparation, including liver function supplements, within 1 week prior to the first administration
10. Individuals with a history of substance abuse or test positive for drugs of abuse on a urine screening test
11. Individuals who had been administered investigational product from other clinical study within the 6 months prior to the first administration
12. Individuals who donated whole blood within the 8 weeks, or blood components within 2 weeks or had a blood transfusion within 4 weeks prior to the first administration of investigational product
13. Woman who are pregnant or breastfeeding
14. Individuals who have difficulty abstaining from omega-3-containing foods(such as oily fish, chia seeds, flaxseeds, walnuts, etc.) from 7 days before the first administration until the end of study
15. Individuals who determines that the tester is unfit to participate in the clinical trial in the final inclusion/exclusion criteria determined by combining the results of the clinical laboratory test conducted on the hospitalization date(-7D)
16. Those who are deemed insufficient to participate in this clinical study by investigators

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss of D352(Part 1) | 1~7day 0 hour, 7day 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hour, 19~21day 0 hour, 21day 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hour
  Area under the D352 concentration in blood-time curve in steady-state
AUCtau,ss of D794(Part 2) | 1day -24 hour~-12 hour, 1~14day 0 hour, 14day 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hour, 19~21day 0 hour, 21day 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hour
  Area under the D794 concentration in blood-time curve in steady-state
Cmax,ss of D352(Part 1) | 1~7day 0 hour, 7day 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hour, 19~21day 0 hour, 21day 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hour
  The maximum D352 concentration in steady-state
Cmax,ss of D794(Part 2) | 1day -24 hour~-12 hour, 1~14day 0 hour, 14day 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hour, 19~21day 0 hour, 21day 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hour
  The maximum D794 concentration in steady-state

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Gwanak-gu, Seoul, South Korea